CLINICAL TRIAL: NCT06175975
Title: The Effect of Auricular Position on Measurement Values and Comfort in Measuring Body Temperature by Tympanic Method in Pediatric Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Hilal Yilmaz, Master's degree student of Fundamentals of Nursing, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IUC-Hyilmaz-001
Record Dates: First submitted 2023-08-06; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Body Temperature Changes
Keywords: Auricular position; Comfort; Pediatric patients
MeSH Terms: conditions — Body Temperature Changes | interventions — methyl hydroxyethyl cellulose

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricular position (Experimental): Experimental group: We will position the auricula back and up first while taking body temperature in pediatric patients. And then we will take body temperature without positioning.
  Interventions: Other: The effect of placing the auricle position on the measurement values and comfort in measurements made with a tympanic membrane thermometer
- Without auricular position (No Intervention): Controlled group: We will not position the auricula first while taking body temperature. And then we will position the auricula back and up.

INTERVENTIONS:
Other: The effect of placing the auricle position on the measurement values and comfort in measurements made with a tympanic membrane thermometer — The effect of placing the auricle position on the measurement values and comfort in measurements made with a tympanic membrane thermometer
  Arms: Auricular position

SUMMARY:
The focus of the clinical research is to examine whether there is a difference in body temperature measurements with or without positioning the auricle in the measurements made with a tympanic membrane thermometer in pediatric patients aged 3-17, and to examine the effect of positioning the ear on comfort behaviors.

DETAILED DESCRIPTION:
It is the nurses' responsibility to monitor vital signs including body temperature, pulse, respiration and blood pressure. Ideal body temperature measurement; It should be a method that is reliable, easy, fast, low-cost, best showing the internal temperature of the body and least affected by environmental conditions. Measurement by the tympanic route; It is a method that is frequently preferred because it gives the correct value, measures the internal temperature, and is not affected by oral nutrition and fluid intake. While the measurement in a few seconds saves nurses time, it is also stated that it is more comfortable for patients than other thermometers.Tympanic membrane thermometers measure the temperature of the blood passing through the tympanic membrane in the ear with infrared radiation.If the tip of the thermometer cannot see the tympanic membrane (eardrum), erroneous results may occur. For this reason, the pinna position where the tip of the tympanic thermometer is placed is very important. It has been stated that in pediatric patients, due to the anatomical structure difference compared to adult patients, measurements should be made by placing them in a downward position. In studies conducted with children and newborns, there are different results in the evidence regarding the effect of auricular position on the measurement value. For this reason, this research is planned to determine the effect of auricular position on body temperature measurement values and comfort behaviors by using Visual Analogue Scale (VAS) and age-appropriate Comfort Daisies developed by Katharine Kolcaba in measurements made with a tympanic membrane thermometer in pediatric patients aged 3-17 years. With the results obtained from this study, it will be evaluated how the auricle position affects the measurement values and comfort behaviors in measuring body temperature by tympanic way in pediatric patients aged 3-17 years. It is thought that the results of this study will contribute to nursing practices and research.

Hypotheses:

H0: There is no significant difference between the body temperature measurement value, VAS score and comfort score performed without pulling the auricle, and the body temperature measurement value, VAS score and comfort score performed by pulling the auricle.

H1: There is a significant difference between the comfort behavior score in the measurement made without pulling the auricle and the comfort behavior score in the measurement made by pulling the auricle.

H2: There is a significant difference between the body temperature measurement value made without pulling the auricle and the body temperature measurement value made by pulling the auricle in patients.

Comparison Hypothesis:

H0: The body temperature measurement value without pulling the auricle, the body temperature measurement value made by pulling the auricle, the VAS score and the comfort score do not differ significantly according to socio-demographic characteristics (age, gender, etc.) and environment.

H1: In patients, the body temperature measurement value without pulling the auricle, the body temperature measurement value made by pulling the auricle, the VAS score and the comfort score show significant differences according to socio-demographic characteristics (age, gender, etc.) and environment.

ELIGIBILITY:
Inclusion Criteria:

1. Being between the ages of 3-17
2. Receiving inpatient care/treatment in the Pediatric Intensive Care Clinic
3. For the pediatric patient, the parents' willingness to participate in the study

Exclusion Criteria:

1. Being outside the age range of 3-17
2. Patient's medical condition;

   * Being sedated or unconscious,
   * Being intubated or tracheostomized,
   * Have had a head injury,
   * Have an ear disease, have an trauma/surgery,
   * Have an ear discharge, ear infection,
   * Have sepsis.
3. Implementation of interventions/treatments that will affect the measurement;

   * Application of treatment (drops) by ear,
   * Last antipyretic treatment taken before 4 hours,
   * Before and during body temperature measurement, interventions (hot and cold application, blood transfusion, hemodialysis and plasma exchange) that will affect the measurement

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-03-22 (Estimated); Study Completion 2024-03-22 (Estimated)

PRIMARY OUTCOMES:
Body temperature changes with or without positioning the auricula in pediatric patients. | 2 minutes
  We will measure the body temperature with tympanic thermometer and will use the Celcius as a measure of unit.
Level of comfort changes (by using Comfort Daisies) with or without positioning the auricula in pediatric patients. | 2 minutes
  We will use Comfort Daisies. Comfort Daisies has 4 daisies which include the expressions like "very good, sort of good, sort of bad and very bad".
Level of comfort changes (by using Visual Analogue Scale) with or without positioning the auricula in pediatric patients. | 2 minutes
  We will use VAS (Visual Analogue Scale).Visual Analogue Scale is between 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal Yilmaz, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Avcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Oguz F, Yildiz I, Varkal MA, Hizli Z, Toprak S, Kaymakci K, Saygili SK, Kilic A, Unuvar E. Axillary and Tympanic Temperature Measurement in Children and Normal Values for Ages. Pediatr Emerg Care. 2018 Mar;34(3):169-173. doi: 10.1097/PEC.0000000000000693. PMID 27050739
- [Result] Uslu S, Ozdemir H, Bulbul A, Comert S, Bolat F, Can E, Nuhoglu A. A comparison of different methods of temperature measurements in sick newborns. J Trop Pediatr. 2011 Dec;57(6):418-23. doi: 10.1093/tropej/fmq120. Epub 2011 Jan 18. PMID 21245075
- [Result] Dante A, Franconi I, Marucci AR, Alfes CM, Lancia L. Evaluating the Interchangeability of Forehead, Tympanic, and Axillary Thermometers in Italian Paediatric Clinical Settings: Results of a Multicentre Observational Study. J Pediatr Nurs. 2020 May-Jun;52:e21-e25. doi: 10.1016/j.pedn.2019.11.014. Epub 2019 Dec 14. PMID 31848034
- [Result] Allegaert K, Casteels K, van Gorp I, Bogaert G. Tympanic, infrared skin, and temporal artery scan thermometers compared with rectal measurement in children: a real-life assessment. Curr Ther Res Clin Exp. 2014 May 8;76:34-8. doi: 10.1016/j.curtheres.2013.11.005. eCollection 2014 Dec. PMID 25067984
- [Result] Kolcaba K, DiMarco MA. Comfort Theory and its application to pediatric nursing. Pediatr Nurs. 2005 May-Jun;31(3):187-94. PMID 16060582
- [Result] Kocoglu H, Goksu S, Isik M, Akturk Z, Bayazit YA. Infrared tympanic thermometer can accurately measure the body temperature in children in an emergency room setting. Int J Pediatr Otorhinolaryngol. 2002 Aug 1;65(1):39-43. doi: 10.1016/s0165-5876(02)00129-5. PMID 12127221
- [Result] Kolcaba KY. A taxonomic structure for the concept comfort. Image J Nurs Sch. 1991 Winter;23(4):237-40. doi: 10.1111/j.1547-5069.1991.tb00678.x. PMID 1937522
- [Result] Kolcaba KY. A theory of holistic comfort for nursing. J Adv Nurs. 1994 Jun;19(6):1178-84. doi: 10.1111/j.1365-2648.1994.tb01202.x. PMID 7930099
- [Result] Childs C, Harrison R, Hodkinson C. Tympanic membrane temperature as a measure of core temperature. Arch Dis Child. 1999 Mar;80(3):262-6. doi: 10.1136/adc.80.3.262. PMID 10325708
- [Result] Pransky SM. The impact of technique and conditions of the tympanic membrane upon infrared tympanic thermometry. Clin Pediatr (Phila). 1991 Apr;30(4 Suppl):50-2; discussion 60. doi: 10.1177/0009922891030004S15. No abstract available. PMID 2029821
- [Result] Orkun N, Eser I. The Effect of Pinna Position on Body Temperature Measurements Made with a Tympanic MembraneThermometer in Pediatric Patients. J Pediatr Res. 2020;7(2):132-8.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT06175975/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT06175975/ICF_001.pdf